CLINICAL TRIAL: NCT02170740
Title: Bioavailability of BIBR 953 ZW After Multiple Oral Doses of 50 and 200 mg BIBR 1048 MS Film-coated Tablet Administered BIDfor 3 Days or 200 mg BIBR 1048 MS With and Without Pre-treatment With Pantoprazole to Healthy Volunteer Subjects. Two Groups, 2-way Crossover, Randomised, Open Trial
Brief Title: Assessment of Safety, Pharmacokinetics and the Effect of BIBR 1048 MS on Coagulation Parameters in Healthy Volunteer Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1160.14
Record Dates: First submitted 2014-06-20; First posted 2014-06-23 (Estimated); Last update posted 2014-06-23 (Estimated); Status verified 2014-06

CONDITIONS: Healthy
MeSH Terms: interventions — Pantoprazole

ARMS (2):
- BIBR 1048 MS (Experimental)
  Interventions: Drug: BIBR 1048 MS - low dose; Drug: BIBR 1048 MS - high dose
- BIBR 1048 MS + Pantoprazole (Experimental)
  Interventions: Drug: BIBR 1048 MS - high dose; Drug: BIBR 1048 MS + Pantoprazole

INTERVENTIONS:
Drug: BIBR 1048 MS - low dose
  Arms: BIBR 1048 MS
Drug: BIBR 1048 MS - high dose
Drug: BIBR 1048 MS + Pantoprazole
  Arms: BIBR 1048 MS + Pantoprazole

SUMMARY:
To assess safety, pharmacokinetics and the effect of BIBR 1048 MS on coagulation parameters in healthy volunteer subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects as determined by results of screening
* Signed written informed consent in accordance with GCP and local legislation
* Age ≥ 18 and ≤ 50 years
* Broca ≥ - 20% and ≤ + 20%

Exclusion Criteria:

* Any finding of the medical examination (including blood pressure, pulse rate and electrocardiogram (ECG)) deviating from normal and of clinical relevance
* History or current gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunologic, hormonal disorders
* History of orthostatic hypotension, fainting spells and blackouts
* Diseases of the central nervous system (such as epilepsy) or psychiatric disorders
* Chronic or relevant acute infections
* History of allergy/hypersensitivity (including drug allergy) which is deemed relevant to the trial as judged by the investigator
* History of any bleeding disorder including prolonged or habitual bleeding
* History of other hematologic disease
* History of cerebral bleeding (e.g. after a car accident)
* History of commotio cerebri
* Intake of drugs with a long-life (> 24 hours) within 1 month prior to administration
* Use of any drug which might influence the results of the trial within 10 days prior to administration or during the trial
* Participation in another trial with investigational drug within 2 months prior to administration or during the trial
* Smoker (> 10 cigarettes or 3 cigars or 3 pipes/day) or inability to refrain from smoking on study days
* Alcohol abuse (> 60g/day)
* Drug abuse
* Blood donation within 1 month prior to administration or during the trial
* Excessive physical activities within 5 days prior to administration or during the trial
* Any laboratory value outside the clinically accepted reference range
* History of any familiar bleeding disorder
* Thrombocytes < 150000/µl

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 1999-11; Primary Completion 2000-01 (Actual)

PRIMARY OUTCOMES:
Urinary excretion of total BIBR 953 ZW | Day 1, day 2, day 3 (different time points)
Peak (maximum) plasma concentration at steady state (Cmax,ss) of BIBR 953 ZW | Day 1, day 2, day 3 (different time points)
Area under the plasma concentration-time curve at steady state (AUCss) of BIBR 953 ZW | Day 1, day 2, day 3 (different time points)
Amount of total (free and glucuronide) BIBR 953 ZW excreted in urine over one dosing interval | Day 1, day 2, day 3 (different time points)

SECONDARY OUTCOMES:
Time to reach the peak plasma concentration (Tmax,ss) of BIBR 953ZW | Day 1, day 2, day 3 (different time points)
Total clearance (CLtot /f ) of BIBR 953 ZW after oral administration | Day 1, day 2, day 3 (different time points)
Occurence of adverse events | 6 weeks
Change from Baseline in pulse rate | Baseline, day 1,day 2, day 3, day 4
Change from Baseline in systolic and diastolic blood pressure | Baseline, day 1,day 2, day 3, day 4
Change from Baseline in clinical laboratory tests | Baseline, day 1,day 2, day 3, day 4
Changes from baseline in activated partial thromboplastin time (aPTT) | Day 1, day 2, day 3 (different time points)
Changes from baseline in prothrombin time (PT) (International Normalised Ratio (INR)) | Day 1, day 2, day 3 (different time points)
Total mean residence time (MRTtot) of BIBR 953 ZW after oral administration | ay 1, day 2, day 3 (different time points)